CLINICAL TRIAL: NCT05051631
Title: BRAVE Strategy - Breast Cancer Risk Assessment -achieVing Equity
Acronym: BRAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Lucy Spalluto, Associate Professor of Radiology and Radiological Sciences, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 211753
Record Dates: First submitted 2021-09-10; First posted 2021-09-21 (Actual); Results first posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: breast cancer; mammogram; screening; risk assessment
MeSH Terms: conditions — Breast Neoplasms | interventions — Methods; Maintenance

STUDY DESIGN:
Intervention Model Description: Stepped-Wedge Trial. 10 clinics will be assigned to 5 arms to receive the intervention at sequential times. The time at which each arm receives the intervention will be randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Intervention plus 12 months maintenance (Experimental): Clinics in this group will be in the control phase for 2 months, receive the 4 month intervention, and be in the maintenance phase for 12 months.
  Interventions: Other: Intervention plus 12 months maintenance
- Intervention plus 10 months maintenance (Experimental): Clinics in this group will be in the control phase for 4 months, receive the 4 month intervention, and be in the maintenance phase for 10 months.
  Interventions: Other: Intervention plus 10 months maintenance
- Intervention plus 8 months maintenance (Experimental): Clinics in this group will be in the control phase for 6 months, receive the 4 month intervention, and be in the maintenance phase for 8 months.
  Interventions: Other: Intervention plus 8 months maintenance
- Intervention plus 6 months maintenance (Experimental): Clinics in this group will be in the control phase for 8 months, receive the 4 month intervention, and be in the maintenance phase for 6 months.
  Interventions: Other: Intervention plus 6 months maintenance
- Intervention plus 4 months maintenance (Experimental): Clinics in this group will be in the control phase for 10 months, receive the 4 month intervention, and be in the maintenance phase for 4 months.
  Interventions: Other: Intervention plus 4 months maintenance

INTERVENTIONS:
Other: Intervention plus 12 months maintenance — The intervention will include 2 months of data collection in the control period, 4 months of education and awareness training, and 12 months of data collection in the maintenance time period.
  Arms: Intervention plus 12 months maintenance
Other: Intervention plus 10 months maintenance — The intervention will include 4 months of data collection in the control period, 4 months of education and awareness training, and 10 months of data collection in the maintenance time period.
  Arms: Intervention plus 10 months maintenance
Other: Intervention plus 8 months maintenance — The intervention will include 6 months of data collection in the control period, 4 months of education and awareness training, and 8 months of data collection in the maintenance time period.
  Arms: Intervention plus 8 months maintenance
Other: Intervention plus 6 months maintenance — The intervention will include 8 months of data collection in the control period, 4 months of education and awareness training, and 6 months of data collection in the maintenance time period.
  Arms: Intervention plus 6 months maintenance
Other: Intervention plus 4 months maintenance — The intervention will include 10 months of data collection in the control period, 4 months of education and awareness training, and 4 months of data collection in the maintenance time period.
  Arms: Intervention plus 4 months maintenance

SUMMARY:
The central goal of this study is to test strategies to implement evidence-based breast cancer risk assessment in healthcare clinics in Tennessee. The BRAVE Strategy (Breast cancer Risk Assessment - achieVing Equity) study aims to assess the feasibility, reach, acceptability, and appropriateness of select customized strategies to increase uptake of breast cancer risk assessment. The investigators will achieve these aims through a conducting a stepped-wedge trial conducted in 10 healthcare clinics in the state of Tennessee. The primary outcome is the proportion of women age 25-49 having risk assessment. Secondary outcomes include the numbers of 1) women identified as high-risk; 2) pursuing risk-adherent screening; and 3) diagnosed with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* ages 25-49

Exclusion Criteria:

* personal history of breast cancer

Ages: 25 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Designated female at birth.
Enrollment: 1071 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucy B Spalluto, MD MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Control: Patients meeting eligibility criteria presenting for visit at an enrolled clinic during the time period prior to intervention (during the control time period).
  Intervention: Patients meeting eligibility criteria presenting for visit at an enrolled clinic during the time period of intervention (during the intervention time period).
  Maintenance: Patients meeting eligibility criteria presenting for visit at an enrolled clinic after intervention (during the maintenance time period).
Pre-assignment Details: Only a single clinic was enrolled. This clinic was in Arm 1 - (2 months control, 4 months intervention,12 months maintenance). Due to lack of clinic resources, the clinic was limited to 9 months of data collection in the maintenance time period.
Units Other Than Participants: Clinics
Groups:
- Arm 1: Arm 1 - 2 months control, 4 months intervention, 12 months maintenance (maintenance limited due to 9 months due to lack of clinic resources)
Period: Overall Study
Arm/Group | Arm 1
Started | 1071; 1 Clinics
Control Group | 299; 1 Clinics
Intervention Group | 362; 1 Clinics
Maintenance Group | 410; 1 Clinics
Completed | 1071; 1 Clinics
Not Completed | 0; 0 Clinics

BASELINE CHARACTERISTICS:
Groups:
- Control: Participants in the control group are those meeting eligibility criteria seen at the enrolled clinic during the control time period (the 2 month baseline time period prior to delivery of the intervention).
- Intervention: Participants in the intervention group are those meeting eligibility criteria seen at the enrolled clinic during the intervention time period (the 4 month time period over which the intervention was delivered).
- Maintenance: Participants in the maintenance group are those meeting eligibility criteria seen at the enrolled clinic during the maintenance time period (the 9 month time period after the delivery of the intervention).
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Maintenance | Total
Number analyzed (Participants) | 299 | 362 | 410 | 1071
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (7.31) | 37.8 (7.55) | 36.6 (7.25) | 37.7 (7.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 299 | 362 | 410 | 1071
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 113 | 132 | 192 | 437
  Ethnicity: Not Hispanic or Latino | 79 | 92 | 75 | 246
  Ethnicity: Unknown or Not Reported | 107 | 138 | 143 | 388
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/Black | 22 | 31 | 33 | 86
  Asian | 1 | 6 | 4 | 11
  American Indian or Alaska Native | 4 | 0 | 17 | 21
  White | 96 | 117 | 82 | 295
  Unknown/Not Reported | 176 | 207 | 270 | 653
  Native Hawaiian/Pacific Islander | 0 | 1 | 0 | 1
  More than once race | 0 | 0 | 4 | 4
Region of Enrollment [Number; unit: participants]
  United States | 299 | 362 | 410 | 1071

OUTCOME MEASURES:

1. Primary Outcome: Number of Eligible Women Who Received Breast Cancer Risk Assessment
Description: The number of women eligible for risk assessment who received documented breast cancer risk assessment.
Time Frame: Baseline (2-months prior to intervention) to 9 months post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention | Maintenance
Number analyzed (Participants) | 299 | 362 | 410
Participants | 8 | 56 | 29

2. Secondary Outcome: Number of Women Who Received Risk Assessment Who Were Identified as High Risk for Breast Cancer.
Description: Number of women who received risk assessment who were identified as high risk for breast cancer. Women are considered high risk if they have 20% or greater lifetime risk of breast cancer using the Tyrer Cuzick risk assessment tool. The Tyrer Cuzick risk assessment tool is an 11 question electronic risk assessment tool about a woman's family history of cancer and personal history to immediately calculate a lifetime risk percentage.
Time Frame: Baseline (2-months prior to intervention) to 9 months post-intervention
Population: For this measure, the denominator includes women who had risk assessment completed and documented.
Measure: Count of Participants; unit: Participants
Groups:
- Control Group: Participants in the control group are those meeting eligibility criteria seen at the enrolled clinic during the control time period (the 2 month baseline time period prior to delivery of the intervention). For this measure, the denominator includes only those who had risk assessment completed.
- Intervention Group: Participants in the intervention group are those meeting eligibility criteria seen at the enrolled clinic during the intervention time period (the 4 month time period over which the intervention was delivered). For this measure, the denominator includes only those who had risk assessment completed.
- Maintenance Group: Participants in the maintenance group are those meeting eligibility criteria seen at the enrolled clinic during the maintenance time period (the 9 month time period after the delivery of the intervention). For this measure, the denominator includes only those who had risk assessment completed.
Arm/Group | Control Group | Intervention Group | Maintenance Group
Number analyzed (Participants) | 8 | 56 | 29
Participants | 0 | 3 | 4

3. Secondary Outcome: Number of Women Identified as High Risk Women Who Received Breast Cancer Screening.
Description: Screening is defined as screening mammography or breast MRI. The number of women who received screening will be identified through from electronic health record review. For this measure, the denominator includes only those who were identified as high risk.
Time Frame: Baseline (2-months prior to intervention) to 9 months post-intervention
Population: For this measure, the denominator includes only those who were identified as high risk.
Measure: Count of Participants; unit: Participants
Groups:
- Control Group: Participants in the control group are those meeting eligibility criteria seen at the enrolled clinic during the control time period (the 2 month baseline time period prior to delivery of the intervention). For this measure, the denominator includes only those who were identified as high risk.
- Intervention Group: Participants in the intervention group are those meeting eligibility criteria seen at the enrolled clinic during the intervention time period (the 4 month time period over which the intervention was delivered). For this measure, the denominator includes only those who were identified as high risk.
- Maintenance Group: Participants in the maintenance group are those meeting eligibility criteria seen at the enrolled clinic during the maintenance time period (the 9 month time period after the delivery of the intervention). For this measure, the denominator includes only those who were identified as high risk.
Arm/Group | Control Group | Intervention Group | Maintenance Group
Number analyzed (Participants) | 0 | 3 | 4
Participants | 0 | 2 | 2

4. Secondary Outcome: Number of Cancers Detected in Women Identified at High Risk.
Description: Cancers will include invasive cancers and cancer in situ. Cancers will be identified from electronic health records. For this measure, the denominator includes only those who were identified as high risk.
Time Frame: Baseline (2-months prior to intervention) to 9 months post-intervention
Population: For this measure, the denominator includes only those who were identified as high risk.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention Group | Maintenance Group
Number analyzed (Participants) | 0 | 3 | 4
Participants | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Baseline (2-months prior to intervention) to 9 months post-intervention
Groups:
- Control Group: Participants in the control group are those meeting eligibility criteria seen at the enrolled clinic during the control time period.
- Intervention Group: Participants in the intervention group are those meeting eligibility criteria seen at the enrolled clinic during the intervention time period.
- Maintenance Group: Participants in the maintenance group are those meeting eligibility criteria seen at the enrolled clinic during the maintenance time period.
Arm/Group | Control Group | Intervention Group | Maintenance Group
All-Cause Mortality (participants affected / at risk) | 0/299 | 0/362 | 0/410
Serious Adverse Events (participants affected / at risk) | 0/299 | 0/362 | 0/410
Other Adverse Events (participants affected / at risk) | 0/299 | 0/362 | 0/410

LIMITATIONS AND CAVEATS:
We had significant difficulty enrolling community clinics during this trial due to the impacts of the COVID 19 pandemic and resulting limitations in clinic resources.

We enrolled a single clinic. This clinic was in Arm 1 - (2 months control, 4 months intervention,12 months maintenance). Due to clinic limited resources, we were also limited to 9 months of data collection in the maintenance time period, rather than the full 12 months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/31/NCT05051631/Prot_SAP_000.pdf